CLINICAL TRIAL: NCT03222661
Title: Direct Comparison of SVOne Obtained Refraction to Subjective Manifest Refraction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Smart Vision Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: SVOne01
Record Dates: First submitted 2017-07-10; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors | interventions — Refraction, Ocular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Refraction — Refractive error measurement

SUMMARY:
The purpose of the study is to compare the final glasses prescription based on refraction obtained with SVOne device to the final prescription obtained via subjective manifest refraction.

DETAILED DESCRIPTION:
Uncorrected refractive error is the leading cause of vision impairment and the second leading cause of blindness worldwide, affecting 1 in 90 individuals (1). In the US population approximately 14 million individuals aged 12 years or older have visual impairment (defined as distance visual acuity of 20/50 or worse), of which more than 11 million individuals (2) could have their vision improved to 20/40 or better with refractive correction.

Uncorrected refractive error impacts all aspects of life, including, but not limited to, loss of employment opportunities, inability to care for family, and inability to receive an education. SVOne is smartphone-based autorefractor, powered by wavefront aberrometry, due to its portability and accuracy it presents as an effective and accessible method of detecting refractive error and dispensing spectacles for better vision (3).

In this study, for each patient, a single clinician will determine final prescription through manifest refraction, while a different clinician will determine final prescription using SVOne exam protocol. Sphere, cylinder and axis will be converted to power vectors and compared by linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 12 (under 18 with parental consent) years of age and older up to 65 years of age.
* No known ocular pathology from previous clinical exams that may limit best corrected visual acuity.

Exclusion Criteria:

* Refractive error greater than +/- 14.00 diopters, or astigmatism greater than -7.00 diopters.
* Known ocular (corneal, lenticular, vitreal, or retinal) pathology that may limit BCVA.
* Best corrected visual acuity with spectacles of 20/25 or worse.
* Any previous surgical or laser procedures that may limit BCVA
* 11 years of age and younger

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population with refractive error between -14.00 to +14.00 diopter of spherical error and astigmatism up to -7.00 diopters.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Sphere, cylinder and axis measurement for each patient | 4 months
  the outcome includes sphere, cylinder and axis measurement (in diopter) by using both SVOne wave-guided autorefractor and subjective manifest refraction
Comparison of two measurements on the same patient | 4 months
  the outcome will include comparison of two sphere, cylinder and axis measurements (in power vectors) for each patient obtained with SVOne wave-guided autorefractor and subjective manifest refraction.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Rosa Pham & Associates, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Naidoo KS, Leasher J, Bourne RR, Flaxman SR, Jonas JB, Keeffe J, Limburg H, Pesudovs K, Price H, White RA, Wong TY, Taylor HR, Resnikoff S; Vision Loss Expert Group of the Global Burden of Disease Study. Global Vision Impairment and Blindness Due to Uncorrected Refractive Error, 1990-2010. Optom Vis Sci. 2016 Mar;93(3):227-34. doi: 10.1097/OPX.0000000000000796. PMID 26905537
- [Background] Vitale S, Cotch MF, Sperduto RD. Prevalence of visual impairment in the United States. JAMA. 2006 May 10;295(18):2158-63. doi: 10.1001/jama.295.18.2158. PMID 16684986
- [Background] Ciuffreda KJ, Rosenfield M. Evaluation of the SVOne: A Handheld, Smartphone-Based Autorefractor. Optom Vis Sci. 2015 Dec;92(12):1133-9. doi: 10.1097/OPX.0000000000000726. PMID 26540478